CLINICAL TRIAL: NCT02577263
Title: Impact of Adjuvant FOLFOX on Quality of Life and Sensory Neurotoxicity in Patients With Advanced Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 019892
Record Dates: First submitted 2015-09-06; First posted 2015-10-16 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Quality of life assessment — Quality of life and chemotherapy induced neurotoxicity evaluation

SUMMARY:
The primary objective of this trial is to determine the impact of the FOLFOX regimen on quality of life and the incidence of chemotherapy induced neurotoxicity.

DETAILED DESCRIPTION:
Gastric cancer is one of the main cancer-related causes of death in the world. There is more than one standard treatment for non-metastatic advanced disease. Among the therapeutic alternatives there is high level of evidence to recommend surgery followed by chemoradiotherapy or chemotherapy and for perioperative chemotherapy. These strategies have not been compared in adequate powered trials, so there are important regional differences in their use. Postoperative chemotherapy with oxaliplatin based chemotherapy may offer some advantages in limited resource settings, because of its lower logistic requirements and it could be specially useful in centers with high quality surgery. On the other hand one of its most important downsides could be a higher impact on quality of life particularly related to oxaliplatin induced neuropathy which can last long after the end of treatment. This is a prospective observational trial in which after consent subjects are going to be evaluated with the EORTC (European Organization for Research and Treatment of Cancer) questionnaires C30 and CIPN20 during FOLFOX (5-fluorouracil/leucovorin with oxaliplatin) adjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gastric adenocarcinoma
* ECOG (Eastern Cooperative Oncology Group) functional status of 0 or 1
* Treated with surgery with curative intent
* TNM stage II - III or TNM stage I with positives lymph nodes

Exclusion Criteria:

* Surgery with microscopical or macroscopical residual tumour
* Adjuvant chemotherapy refusal
* ECOG functional status of 2 or more
* Previous peripheral neuropathy
* Significant cardiovascular disease or other organ disfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histological diagnosis of gastric adenocarcinoma who were treated with surgery
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2015-04; Primary Completion 2017-01 (Actual); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Quality of life deterioration > 10% (dichotomic) | Participants will be followed until 3 months after the end of chemotherapy for this outcome, an expected average of 9 months
  Questionnaire EORTC C30 (sub scale global health status) in two consecutive evaluation

SECONDARY OUTCOMES:
Disease free survival | Participants will be followed until 2 years after the end of chemotherapy for this outcome, an expected average of 24 months
  Time to event
Overall survival | Participants will be followed until 2 years after the end of chemotherapy for this outcome, an expected average of 24 months
  Time to event
Significant chemotherapy induced neurotoxicity > 10% (dichotomic) | Participants will be followed until 3 months after the end of chemotherapy for this outcome, an expected average of 9 months
  Questionnaire EORTC CIPN20 (sensory sub scale) in two consecutive evaluation
Median change in Quality of life score | Participants will be followed until 3 months after the end of chemotherapy for this outcome, an expected average of 9 months
  Questionnaire EORTC C30
Median change in chemotherapy induced neurotoxicity score | Participants will be followed until 3 months after the end of chemotherapy for this outcome, an expected average of 9 months
  Questionnaire EORTC CIPN20
Quality of life deterioration > 10% | Participants will be followed until 3 months after the end of chemotherapy for this outcome, an expected average of 9 months
  Time to event considering the a drop of 10% in the global health sub scale of the EORTC C30 Questionnaire
Significant chemotherapy induced neurotoxicity > 10% | Participants will be followed until 3 months after the end of chemotherapy for this outcome, an expected average of 9 months
  Time to event considering the a drop of 10% in the sensory sub scale of the EORTC CIPN 20 Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sebastián Mondaca, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Dr. Sótero del Río Hospital, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided